CLINICAL TRIAL: NCT02228460
Title: A Phase 2 Study to Evaluate the Safety, Pharmacodynamics, Pharmacokinetics, and Exploratory Efficacy of GZ/SAR402671 in Enzyme Replacement Therapy (ERT) Treatment-naïve Adult Male Patients Diagnosed With Fabry Disease
Brief Title: Evaluate the Safety, Pharmacodynamics, Pharmacokinetics, and Exploratory Efficacy of GZ/SAR402671 in Treatment-naïve Adult Male Patients With Fabry Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACT13739; 2013-005324-41; U1111-1152-1456 (Other: UTN)
Record Dates: First submitted 2014-08-27; First posted 2014-08-29 (Estimated); Results first posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2016-09

CONDITIONS: Fabry Disease
Keywords: Venglustat
MeSH Terms: conditions — Fabry Disease | interventions — venglustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GZ/SAR402671 (Experimental): GZ/SAR402671 15 milligram (mg) once daily orally for 26 weeks.
  Interventions: Drug: GZ/SAR402671

INTERVENTIONS:
Drug: GZ/SAR402671 — Pharmaceutical form: Capsule; Route of administration: Oral

SUMMARY:
Primary Objective:

To assess the safety, pharmacokinetics (PK), pharmacodynamics (PD), and exploratory efficacy of GZ/SAR402671 in enzyme replacement therapy treatment-naïve adult male participants diagnosed with Fabry disease.

DETAILED DESCRIPTION:
The total duration of study per participant was 7 to 8 months for participants who entered a planned extension study and approximately 13 to 14 months for participants who did not enter a planned extension study. A 2-year extension study was planned for eligible participants.

ELIGIBILITY:
Inclusion criteria:

* The participant was greater than equal to (>=) 18 years of age and less than (<) 50 years of age.
* The participant was male.
* The participant had provided a signed informed consent.
* The participant had a confirmed diagnosis of Fabry disease as documented by leukocyte α- Galactosidase A (αGAL) activity of <4 nanomole/hour/milligram (nmol/hr/mg) leukocyte (preferred assay; results from a central laboratory) or plasma αGAL <1.5 nanomole/hour/milliliter (nmol/hr/mL) (results from a central laboratory).
* The participant had a plasma globotriaosylsphingosine (lyso-GL3) >=65 nanogram per milliliter (ng/mL).
* The participant had never been treated with a Fabry disease-specific treatment.
* If the participant was on renin-angiotensin-aldosterone system (RAAS) blockers and antidepressants, the dose should be stable (i.e., prescribed dose and frequency) for at least the immediate 3 months prior to screening.

Exclusion criteria:

* The participant had an estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m^2 using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI).
* The participant had a median urine protein/creatinine ratio (PCR) >=0.5 gram per gram (g/g) (median of 3 overnight urine collections. Collection of each of the 3 samples must occur between 4 and 7 days of each other, and all samples must be collected within a 15 day period). All 3 samples must be collected regardless of the results and results available prior to Day 1.
* The participant had undergone a kidney transplant.
* The participant had either active or a history of clinically significant organic disease (with the exception of the symptoms related to Fabry disease), including clinically significant cardiovascular, hepatic, pulmonary, hematologic, neurological or renal disease, or other medical condition, serious inter-current illness, or extenuating circumstances that, in the opinion of the Investigator, would preclude participation in the trial.
* The participant had abnormal liver function (serum total bilirubin > the upper limit of normal, or serum alanine aminotransferase ([ALT] and aspartate aminotransferase [AST] >2.0 times the upper limit of normal).
* The participant had, according to World Health Organization (WHO) grading a cortical cataract (COR) > one-quarter of the lens circumference (Grade COR-2) or a posterior subcapsular cataract (PSC) >2 millimeter (mm) (Grade PSC-2). Participants with nuclear cataracts were not excluded.
* The participant was currently receiving potentially cataractogenic medications.
* The participant had received strong or moderate inducers or inhibitors of Cytochrome P450 3A4 (CYP3A4) per Food and Drug Administration (FDA) classification within 14 days prior to enrollment or within 5 times the elimination half-life or PD half-life of the medication, whichever is longer.
* The participant was scheduled for in-patient hospitalization, including elective surgery, during the study.
* The participant had a positive result on any of the following tests: hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti-HIV2 Ab). Participants with a positive hepatitis B surface antibody (HBsAb) test with a history of prior hepatitis B immunization were eligible if other criteria met (i.e., negative tests for: HBsAg, hepatitis B core antibody [HBcAb], and hepatitis C virus antibody [HCVAb]).
* The participant had participated in a study involving an investigational drug within the past 30 days of the start of the trial.
* The participant was unwilling to comply with the requirements of the protocol.
* The participant was a sexually active man who was not willing to use 2 forms of birth control including a barrier method during the study until 6 weeks after the last treatment with investigational medicinal product (IMP).
* The participant had a history or ongoing clinically significant cardiac arrhythmia, defined as either atrial fibrillation, sustained or non-sustained ventricular tachycardia.
* The participant had any contraindication to magnetic resonance imaging (MRI).
* The participant had one of the following central nervous system exclusion criteria:

  * Acute stroke, within 3 months of the screening visit.
  * History of seizures.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (8):
- United States (3):
  - Investigational Site Number 840002, Atlanta, Georgia
  - Investigational Site Number 840003, Cincinnati, Ohio
  - Investigational Site Number 840001, Fairfax, Virginia
- Investigational Site Number 250001, Garches, France
- Investigational Site Number 616001, Warsaw, Poland
- Investigational Site Number 643002, Moscow, Russia
- United Kingdom (2):
  - Investigational Site Number 826003, Birmingham
  - Investigational Site Number 826002, Cambridge

REFERENCES:
- [Derived] Deegan PB, Goker-Alpan O, Geberhiwot T, Hopkin RJ, Lukina E, Tylki-Szymanska A, Zaher A, Sensinger C, Gaemers SJM, Modur V, Thurberg BL, Sharma J, Najafian B, Mauer M, DasMahapatra P, Wilcox WR, Germain DP. Venglustat, an orally administered glucosylceramide synthase inhibitor: Assessment over 3 years in adult males with classic Fabry disease in an open-label phase 2 study and its extension study. Mol Genet Metab. 2023 Feb;138(2):106963. doi: 10.1016/j.ymgme.2022.11.002. Epub 2022 Nov 9. PMID 36481125

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study at 8 centers in 5 countries between 11 November 2014 and 06 September 2016. A total of 14 participants were screened in the study.
Pre-assignment Details: Out of 14 screened participants, 11 participants were enrolled and treated in the study.
Groups:
- GZ/SAR402671: GZ/SAR402671 15 milligram (mg) once daily, orally for 26 weeks.
Period: Overall Study
Arm/Group | GZ/SAR402671
Started | 11
Completed | 9
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on full analysis set (FAS) that included all participants who received at least 1 dose of study treatment.
Groups:
- GZ/SAR402671: GZ/SAR402671 15 mg once daily, orally for 26 weeks.
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.5 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Week 26 in Skin Globotriaosylceramide (GL-3) Score in Superficial Skin Capillary Endothelium: Number of Participants in Categories of Shift in GL-3 Score From Baseline to Week 26
Description: Skin biopsies taken at Baseline and Week 26 were analyzed for cellular GL-3 accumulation (inclusions) by light microscopy. Three independent pathologists evaluated each biopsy using an inclusion severity score of 0 (none/trace), 1 (mild), 2 (moderate), and 3 (severe), where higher score indicated more severe condition. A single score per participant per time point was derived by taking the score rated by a majority of the pathologists; if a majority score could not be derived, the median score was used. Data were summarized and reported in terms of number of participants with shift from Baseline GL-3 score to Week 26 GL-3 score. Any shift category of Baseline score/Week 26 score that was not observed is not reported. Shift to lower score from Baseline to Week 26 indicates less severe condition at Week 26.
Time Frame: Baseline, Week 26
Population: Analysis was performed on full analysis set (FAS) that included all participants who received at least 1 dose of study treatment. Here, 'overall number of participants analyzed' = participants with available data at both Baseline and Week 26.
Measure: Count of Participants; unit: Participants
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 9
Participants
  Baseline Score: 1 / Week 26 Score: 1 | 4
  Baseline Score: 1 / Week 26 Score: 2 | 1
  Baseline Score: 2 / Week 26 Score: 1 | 3
  Baseline Score: 2 / Week 26 Score: 2 | 1
Statistical Analysis 1: Comparison: GZ/SAR402671; A McNemar test was used to test the treatment effect based on paired pre-treatment and post-treatment (Week 26) frequencies of skin GL-3 score grouped into the categories (0 to <2; 2 to 3); Test type: Other; p = 0.3173, McNemar Test — Threshold for significance at 0.05 level

2. Primary Outcome: Mean Change From Baseline at Week 26 in Skin GL-3 Score in Superficial Skin Capillary Endothelium
Description: Skin biopsies taken at Baseline and Week 26 were analyzed for cellular GL-3 accumulation (inclusions) by light microscopy. Three independent pathologists evaluated each biopsy using an inclusion severity score of 0 (none/trace), 1 (mild), 2 (moderate), and 3 (severe), where higher score indicated more severe condition. A single score per participant per time point was derived by taking the score rated by a majority of the pathologists; if a majority score could not be derived, the median score was used. Change from Baseline in GL-3 score was obtained by subtracting Baseline value from post-baseline value at Week 26. A negative change from Baseline indicates less severe condition at Week 26.
Time Frame: Baseline, Week 26
Population: Analysis was performed on FAS. Here, 'overall number of participants analyzed' = participants with available data at both Baseline and Week 26.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 9
score on a scale | -0.22 [-0.73 to 0.29]
Statistical Analysis 1: Comparison: GZ/SAR402671; Wilcoxon signed rank test was used to assess the mean change from Baseline to Week 26 in skin GL-3 score; Test type: Other; p = 0.625, Wilcoxon signed rank test — Threshold for significance at 0.05 level

3. Secondary Outcome: Change From Baseline in Plasma GL-3 Concentration at Week 26
Description: Change from Baseline in plasma GL-3 was obtained by subtracting Baseline value from post-baseline value at Week 26. Concentration of GL-3 in plasma was determined using a validated liquid chromatography tandem mass spectrometry (LC-MS/MS) method.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 9
mcg/mL | -3.62 (1.07)

4. Secondary Outcome: Change From Baseline in Plasma Lyso Globotriaosylceramide (Lyso-GL-3) Concentration at Week 26
Description: Change from Baseline in plasma Lyso-GL-3 was obtained by subtracting Baseline value from post-baseline value at Week 26. Concentration of lyso-GL-3 in plasma was determined using a validated LC-MS/MS method.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 9
ng/mL | -30.99 (22.83)

5. Secondary Outcome: Change From Baseline in Plasma Glucosylceramide (GL-1) Concentration at Week 26
Description: Change from Baseline in plasma GL-1 was obtained by subtracting Baseline value from post-baseline value at Week 26. Concentration of GL-1 in plasma was determined using a validated LC-MS/MS method.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 9
mcg/mL | -3.26 (1.43)

6. Secondary Outcome: Change From Baseline at Week 26 in Skin GL-3 Score in Deep Vessels Endothelial Cells: Number of Participants in Categories of Shift in GL-3 Score From Baseline to Week 26
Description: as for outcome 1
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 9
Participants
  Baseline Score: 1 / Week 26 Score: 1 | 1
  Baseline Score: 2 / Week 26 Score: 1 | 2
  Baseline Score: 2 / Week 26 Score: 2 | 6

7. Secondary Outcome: Change From Baseline at Week 26 in Skin GL-3 Score in Deep Vessels Smooth Muscle Cells: Number of Participants in Categories of Shift in GL-3 Score From Baseline to Week 26
Description: as for outcome 1
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 9
Participants
  Baseline Score: 1.5 / Week 26 Score: 1.5 | 2
  Baseline Score: 2 / Week 26 Score: 2 | 7

8. Secondary Outcome: Change From Baseline at Week 26 in Skin GL-3 Score in Perineurium Cells: Number of Participants in Categories of Shift in GL-3 Score From Baseline to Week 26
Description: as for outcome 1
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 9
Participants
  Baseline Score: 1 / Week 26 Score: 2 | 1
  Baseline Score: 2 / Week 26 Score: 2 | 8

9. Secondary Outcome: Change From Baseline in Urine Globotriaosylceramide (GL-3) Concentration at Week 26
Description: Change from Baseline in urine GL-3 was obtained by subtracting Baseline value from post-baseline value at Week 26. Concentration of GL-3 in urine was determined using a validated LC-MS/MS method.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/mmol Cr
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 8
mg/mmol Cr | -0.25 (0.19)

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Any untoward medical occurrence in a participant who received study drug was considered an adverse event (AE) without regard to possibility of causal relationship with this treatment. TEAEs were defined as AEs that developed or worsened during on-treatment period (period from the first administration of study drug through the last administration of the study drug plus 30 days or end of study participation for participant, whichever occurs first).
Time Frame: From Baseline up to 212 days
Population: Analysis was performed on safety population which included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
Participants | 9

11. Secondary Outcome: Pharmacokinetics (PK): Maximum Plasma Drug Concentration (Cmax) of GZ/SAR402671
Description: Maximum plasma concentration observed for study drug was reported.
Time Frame: Day 1 (predose and 1, 2, 4, 8, and 24 hours post-dose); Day 182 (predose and 1, 2, 4, 8, and 24 hours post-dose)
Population: Analysis was performed on PK population which included all participants for whom the primary PK data were considered sufficient and interpretable. Here, 'number analyzed' = participants with available data at specified time-point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
ng/mL
  Day 1 | 24.7 (5.89)
  Day 182: number analyzed (Participants) | 9
  Day 182 | 192.0 (96.4)

12. Secondary Outcome: PK: Plasma Trough Concentration (Ctrough) of GZ/SAR402671
Description: Ctrough was defined as the plasma concentration of study drug observed just before treatment administration during repeated dosing.
Time Frame: Predose on Days 14, 28, 56, 84, 126, and 182
Population: Analysis was performed on PK population. Here, 'number analyzed' = participants with available data at specified time-point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
ng/mL
  Day 14 | 152.0 (68.9)
  Day 28 | 165.0 (66.1)
  Day 56: number analyzed (Participants) | 10
  Day 56 | 182.0 (90.3)
  Day 84: number analyzed (Participants) | 10
  Day 84 | 164.0 (124.0)
  Day 126: number analyzed (Participants) | 9
  Day 126 | 175.0 (94.7)
  Day 182: number analyzed (Participants) | 9
  Day 182 | 164.0 (89.4)

13. Secondary Outcome: PK: Time to Reach Maximum Plasma Drug Concentration (Tmax) of GZ/SAR402671
Description: Tmax was defined as time to reach maximum plasma concentration of study drug.
Time Frame: Day 1 (predose and 1, 2, 4, 8, and 24 hours post-dose); Day 182 (predose and 1, 2, 4, 8, and 24 hours post-dose)
Population: as for outcome 12
Measure: Median (Full Range); unit: hours
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
hours
  Day 1 | 8.00 [1.07 to 24.00]
  Day 182: number analyzed (Participants) | 9
  Day 182 | 4.00 [0.00 to 8.00]

14. Secondary Outcome: PK: Area Under Plasma Concentration Versus Time Curve From 0 to 24 Hours (AUC0-24) of GZ/SAR402671
Description: Area under the plasma concentration versus time curve of study drug from time 0 to 24 hours (AUC0-24) was calculated using the trapezoidal method over the dosing interval.
Time Frame: Day 1 (predose and 1, 2, 4, 8, and 24 hours post-dose); Day 182 (predose and 1, 2, 4, 8, and 24 hours post-dose)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
ng*hour/mL
  Day 1 | 476 (125)
  Day 182: number analyzed (Participants) | 9
  Day 182 | 4110 (2090)

15. Secondary Outcome: PK: Terminal Half-life (t1/2z) of GZ/SAR402671
Description: Plasma t1/2z was the time measured for the plasma concentration of drug to decrease by one half. The t1/2z was estimated based on 24-hour post-dose PK.
Time Frame: Day 1 (predose and 1, 2, 4, 8, and 24 hours post-dose); Day 182 (predose and 1, 2, 4, 8, and 24 hours post-dose)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 11
hours
  Day 1: number analyzed (Participants) | 4
  Day 1 | 86.8 (39.6)
  Day 182: number analyzed (Participants) | 7
  Day 182 | 128.0 (59.0)

16. Secondary Outcome: PK: Apparent Total Body Clearance of GZ/SAR402671 at Steady State (CLss/F)
Description: Apparent total body clearance at steady state was a quantitative measure of rate of clearance of drug from the blood following oral administration, and is described in terms of volume of fluid clear of drug per time unit (eg, mL/min).
Time Frame: Predose and 1, 2, 4, 8, and 24 hours post-dose on Day 182
Population: Analysis was performed on PK population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: mL/hour
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 9
mL/hour | 7490 (10900)

17. Secondary Outcome: PK: Apparent Volume of Distribution of GZ/SAR402671 (Vss/F) at Steady State
Description: Volume of distribution at steady state was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of drug.
Time Frame: Predose and 1, 2, 4, 8, and 24 hours post-dose on Day 182
Population: Since the percent extrapolation of AUC for all participants was >30%, AUC could not be determined and hence, Vss/F could not be calculated.
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 0

18. Secondary Outcome: PK: Cumulated Amount of GZ/SAR402671 Excreted in Urine From 0 to 24 Hours (Ae0-24)
Description: Ae0-24 was the cumulated amount of study drug excreted in urine during the time interval of 0 to 24 hours.
Time Frame: 0-24 hours on Day 182
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 9
mcg | 3210.0 (1640.0)

19. Secondary Outcome: PK: Percentage of Dose of GZ/SAR402671 Excreted in Urine From 0 to 24 Hours (fe0-24)
Description: fe0-24 was the fraction of dose excreted in urine during the time interval of 0 to 24 hours.
Time Frame: 0-24 hours on Day 182
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percentage of dose
Groups:
- GZ/SAR402671: GZ/SAR402671 15 mg once daily orally for 26 weeks.
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 9
percentage of dose | 21.4 (10.9)

20. Secondary Outcome: PK: Renal Clearance (CLR) of GZ/SAR402671 From 0 to 24 Hours
Description: CLR was calculated by dividing the cumulative amount of drug excreted in urine during the dosing interval of 0-24 hours by area under the plasma drug concentration time-curve during the dosing interval of 0-24 hours.
Time Frame: 0-24 hours on Day 182
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: mL/hour
Arm/Group | GZ/SAR402671
Number analyzed (Participants) | 9
mL/hour | 925 (407)

ADVERSE EVENTS:
Time Frame: Baseline up to 212 days
Description: Reported AEs are TEAEs that is AEs developed/worsened during "on treatment period" (from first administration through last administration of study drug + 30 days or end of study participation for participant, whichever occurs first). Analysis was performed on safety population that included all enrolled participants who received at least 1 dose of study drug.
Arm/Group | GZ/SAR402671
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 3/11
Other Adverse Events (participants affected / at risk) | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GZ/SAR402671 (N=11)
Haemolysis (Blood and lymphatic system disorders) | 1
Floppy infant (Musculoskeletal and connective tissue disorders) | 1
Depressed mood (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GZ/SAR402671 (N=11)
Atrial fibrillation (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 2
Blepharitis (Eye disorders) | 1
Chalazion (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Lenticular opacities (Eye disorders) | 1
Retinal vascular disorder (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Oesophageal discomfort (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 2
Feeling hot (General disorders) | 2
Influenza like illness (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pyrexia (General disorders) | 2
Ear infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Muscle strain (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Electrocardiogram T wave abnormal (Investigations) | 1
Electrocardiogram abnormal (Investigations) | 1
Nuclear magnetic resonance imaging brain abnormal (Investigations) | 1
Vibration test abnormal (Investigations) | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Amnesia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 4
Hypoaesthesia (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Sinus headache (Nervous system disorders) | 1
White matter lesion (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depressed mood (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Angiokeratoma (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.